CLINICAL TRIAL: NCT05683106
Title: Effects of the Use of Customized Silicone Digital Orthoses on Pre-ulcerative Lesions and Plantar Pressure During Walking in People With Diabetic Neuropathy: a Randomized Controlled Clinical Trial
Brief Title: Effects of Customized Silicone Digital Orthoses in People With Diabetic Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Isabel de Camargo Neves Sacco, Associate Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LaBiMPH03
Record Dates: First submitted 2022-12-20; First posted 2023-01-12 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Neuropathies
Keywords: Diabetes Mellitus; Diabetic foot; Plantar pressure; Orthosis digital; quality of life
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The participants will receive a custom silicone digital orthosis (CSDO) to realign the toes according to their needs. They will be instructed to use the CSDO throughout the day, remove it to sleep and reposition it on the foot the next day. Furthermore they will be assisted by a stomatherapy specialist, dermatology or clinical podiatry nurse and will receive foot care for thinning the calluses, referral (if necessary) to the Specialized Rehabilitation Center - CER, health equipment linked to SUS, for the purchase of insoles and/ or molded footwear (when indicated) and guidance on the use of therapeutic footwear.
  Interventions: Device: Custom silicone digital orthosis (CSDO)
- Control Group (No Intervention): The participants will be assisted by the stomatherapy specialist, dermatology or clinical podiatry nurse and will receive foot care for thinning the calluses, referral (if necessary) to the Specialized Rehabilitation Center - CER, health equipment linked to SUS, for the purchase of insoles and/ or molded footwear (when indicated) and guidance on the use of therapeutic footwear.

INTERVENTIONS:
Device: Custom silicone digital orthosis (CSDO) — Custom silicone digital orthosis (CSDO) will be made under mold to provide realignment of toes, protection or replacement of a segment that was amputated.They will be indicated for corrections of rigid/fixed or flexible toes deformities.CSDO will be constructed using different types of silicone and different hardness considering whether the deformities are rigid or flexible and,when necessary,these components of the orthoses will be merged.Intervention participants will be asked to clean the CSDO and interdigital spaces with soap and water;adequate drying of the fingers and interdigital region;always wear the CSDO with appropriate footwear and socks;keep monitoring the integrity of the CSDO and always communicate any identification of changes in the feet or CSDO.Adverse effects will be evaluated, such as:possible skin irritation; discomfort or pain;contractures;trauma due to friction.Adherence will be verified every 3 months and via telephone contact,monthly.
  Arms: Intervention Group

SUMMARY:
The present study aims to evaluate the efficacy and safety of the use of customized silicone digital orthoses for six months in the distribution of plantar pressure, in the reduction of pre-ulcerative lesions and plantar ulcers in the forefoot, foot deformities, quality of life and foot health and functionality in people with diabetes and neuropathy with risk category 2 and 3 for ulcers, according to the International Working Group on Diabetic Foot.

DETAILED DESCRIPTION:
The present study aims to evaluate the effects and safety of the use of customized silicone digital orthoses for six months in the plantar pressure distribution during gait, in the reduction of pre-ulcerative lesions and plantar ulcers at forefoot, in functional balance, foot deformities, quality of life and foot health and functionality in people with diabetes and and diabetic neuropathy with risk category 2 and 3, according to the International Working Group on Diabetic Foot.

The sample will consist of 60 participants, who will be randomly allocated, in a randomized controlled clinical trial, in the control or intervention groups and evaluated at baseline, 3 and 6 months of follow up. The assessment includes (1) classification of the risk of foot ulceration, (2) analysis of plantar pressure during gait, (3) quality of life, (4) foot deformities, (5) pre-ulcerative lesions, (6) functionality and general health of the feet.

The hypothesis of this study is that the intervention group will present a reduction in the peak pressures during gait, a reduction in hyperkeratosis at forefoot, a reduction in the incidence and recurrence of forefoot ulcerations, and improved quality of life and in the functionality and health of the foot, when compared to the control group after six months of use of silicone digital orthoses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed type 1 or 2 diabetes, with diabetic peripheral neuropathy confirmed by loss of sensitivity measured by 10 g Semmes-Weinstein monofilament or 128Hz tuning fork and by the fuzzy score (www.usp.br/labimph/fuzzy);
* Presence of 1 or more deformities at the forefoot region (claw toes, hammer toes, mallet toes, overlapping toes, hallux valgus, prominence of the metatarsal heads or reduction/displacement of the fat pad);
* Ability to walk independently with or without the aid of a walking device;

Exclusion Criteria:

* Presence of other diagnosed neurological diseases;
* Presence of dementia or inability to give consistent information;
* Presence of major vascular complications;
* Receiving any physiotherapy intervention;
* Major vascular complications (ischemia)
* Presence of an active ulcer at the time of baseline assessment;
* Major amputations;
* Minor amputations, except toes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Pre-ulcerative lesions and ulcers at 12 and 24 weeks | 12-weeks, 24-weeks
  It will be evaluated according to a study, which classifies hyperkeratosis into 6 degrees

SECONDARY OUTCOMES:
Change from Baseline Dynamic Plantar Pressure Distribution during gait at 12 and 24 weeks | 12 and 24 weeks
  A pressure platform (emed®-q100, novel, Germany) will be used to assess peak pressure (kPa) in the forefoot region during walking.
Change from Baseline Foot health and functionality at 12 and 24 weeks | 12 and 24 weeks
  The Brazilian version of the Foot-Health Status Questionnaire (FHSQ-BR) will be used. This instrument is divided into three domains and we are using domains I and II. The first domain evaluates the foot in four spheres: pain, function, footwear and general health. The second domain evaluates the general state of health, also in four spheres: general health, physical activity, social capacity and vitality. Domains I and II are composed of questions with answer choices that are presented in the affirmative sentences and corresponding numbers. Domain III, which is not being used, comprises the collection of general demographic data of individuals. Each domain receives a score from 0 to 100, where 100 expresses the best condition and 0 to worst.
Change from baseline of the Quality of life at 12 and 24 weeks | 12 and 24 weeks
  Participants will answer the EQ-5D questionnaire, which is an instrument for measuring health-related quality of life that allows generating an index representing the value of an individual's health status.
Change from Baseline Safety at 12 weeks | 12 weeks
  To assess safety with the use of orthoses, a closed structured questionnaires will be applied, consisting of 11 questions related to safety. Responses will be evaluated using a 5-point Likert scale (1 = strongly agree; 2 = agree; 3 = neither agree nor disagree; 4 = disagree; 5 = strongly disagree).
Change from Baseline Satisfaction at 12 weeks | 12 weeks
  To assess satisfaction with the use of orthoses, a closed structured questionnaires will be applied, consisting of 7 related to satisfaction. Responses will be evaluated using a 5-point Likert scale (1 = strongly agree; 2 = agree; 3 = neither agree nor disagree; 4 = disagree; 5 = strongly disagree).
Change from Baseline Comfort at 12 weeks | 12-weeks
  To assess comfort with the use of orthoses, a Visual Analogue Scale (VAS) will be applied, consisting of 0 and 10 marked points, in which 0 indicates no discomfort and 10 indicates the highest level of discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel C Sacco, PhD, Principal Investigator — Associate Professor at São Paulo University
Locations (1):
- Stay Care Clinica, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lucoveis MLS, Gamba M, Silva EQ, Pinto LAS, Sacco ICN. The effects of the use of customized silicone digital orthoses on pre-ulcerative lesions and plantar pressure during walking in people with diabetic neuropathy: A study protocol for a randomized controlled trial. Contemp Clin Trials Commun. 2023 Dec 23;37:101247. doi: 10.1016/j.conctc.2023.101247. eCollection 2024 Feb. PMID 38269045
- See also: University of Sao Paulo website — http://www.usp.br
- See also: Laboratory of Biomechanics of Human Movement and Posture website — http://www.usp.br/labimph